CLINICAL TRIAL: NCT06850909
Title: Evaluating the Influence of 3D Culture Dish Design on Preimplantation Genetic Development in Sibling Oocytes: a Randomized Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ganin Fertility Center (Other)
Responsible Party: Principal Investigator, Eman Hasanen, ESHRE certified Clinical Embryologist, Ganin Fertility Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFC-0010
Record Dates: First submitted 2025-02-26; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Embryo Culture
Keywords: 3D culture dish; embryo culture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dish no.1 (Active Comparator): Sibling oocytes were randomly allocated for culture in Dish 1 (Microdrop GPS Dish) from the ICSI procedure until the blastocyst stage.
  Interventions: Device: Microdrop GPS dish
- Dish no.2 (Active Comparator): Sibling oocytes were randomly allocated for culture in Dish 1 (16 well BIRR Dish) from the ICSI procedure until the blastocyst stage.
  Interventions: Device: 16 well BIRR dish

INTERVENTIONS:
Device: Microdrop GPS dish — The µDrop GPS® micro-wells dish is specifically designed for oocyte and embryo handling and culture. The sloped concave micro-well bottoms of the µDrop GPS® dish allow oocytes and embryos to settle at a central location away from the well walls. The concave nature of the wells provides the thinnest well bottom possible, helping to reduce refraction and allow for optimal visualization. The wells may reduce droplet collapsing/mixing, offer better orientation/optics, and reduce set-up/observation time.
  Arms: Dish no.1
Device: 16 well BIRR dish — The 16-Well BIRR Dish is a high-quality 3D culture dish designed for optimal embryo handling and identification in IVF. It features well-numbering (1-16) for clear tracking, a large labeling area, and an expanded working space for better accessibility. Its 16 wells allow for increased wash drops and single embryo culture, reducing the number of dishes needed per IVF cycle. Rigorously tested (MEA+, LAL, and SMA per lot), it ensures safe and efficient embryo culture.
  Arms: Dish no.2

SUMMARY:
Evaluating the Influence of 3D Culture Dish Design on Preimplantation Genetic Development in Sibling Oocytes: A Randomized Trial

DETAILED DESCRIPTION:
The configuration of culture dishes plays a crucial role in preimplantation embryo development by influencing key culture conditions such as media distribution, oxygen exchange, and embryo spacing, all of which directly impact embryonic growth, fertilization, blastocyst formation, and overall blastocyst quality. Traditional 2D culture dishes provide a flat surface for embryo development, whereas 3D culture dishes create a microenvironment that better mimics in vivo conditions by optimizing nutrient availability and reducing stress from environmental fluctuations. In this study, we compare the effects of two different 3D culture dishes-Dish 1 (Microdrop GPS Dish) and Dish 2 (16-Well BIRR Dish)-on preimplantation genetic outcomes. Using a sibling oocyte split design, oocytes were randomly divided after intracytoplasmic sperm injection (ICSI) and cultured in either dish, ensuring that each patient serves as their own internal control. Embryo development was closely monitored from fertilization to blastocyst formation, to determine whether dish design has a significant impact on preimplantation embryo development.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 35 years or younger
* A minimum of 15 mature oocytes available for ICSI
* Classified as a good prognosis patient

Exclusion Criteria:

* Cases with severe DNA fragmentation
* Patients undergoing FNA or TESE procedures
* Severe male factor infertility
* History of low or failed fertilization in previous cycles
* Any contraindications to gonadotropin stimulation
* Presence of leukocytospermia

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Blastocyst Development rate | 5 - 6 days
  Defined as the proportion of blastocysts formed on day 5 or 6

SECONDARY OUTCOMES:
Fertilization rate | 1 day
  Defined as the proportion of fertilized oocytes
Cleavage rate | 3 days
  Defined as the proportion of cleaved embryos on day 3
Blastocyst Quality rate | 5 - 6 days
  Defined as the assessment of blastocyst quality according to Gardner's criteria into: good, fair or poor
High Quality Day 3 rate | 3 days
  proportion of high quality day 3 embryos

CONTACTS AND LOCATIONS:
Locations (1):
- Ganin Fertility Center, Cairo, Egypt